CLINICAL TRIAL: NCT06908824
Title: The No Endotamponade for Macular Hole Repair (NEMAR) Study: An International Multi-center Randomized Controlled Trial Comparing Macular Hole Closure Using Internal Limiting Membrane Flap Without Endotamponade Versus Conventional Surgery
Brief Title: No Endotamponade for Macular Hole Repair: the NEMAR Study
Acronym: NEMAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Poznan University of Medical Sciences (Other); Chang Gung University (Other)
Responsible Party: Principal Investigator, Simon KH Szeto, Clinical assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2025-084-2
Record Dates: First submitted 2025-03-24; First posted 2025-04-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Macular Hole; Macular Hole Surgery
Keywords: Macular Hole; Vitrectomy; Macular surgery; Internal limiting membrane peeling; Gas tamponade
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgery (Active Comparator): Patients would undergo conventional surgery to repair macular hole and be instructed to adopt a face-down posturing in the first 5 days following operation.
  Interventions: Procedure: Conventional surgery
- Internal limiting membrane (ILM) flap with no gas tamponade (Experimental): Patients would undergo macular hole repair by the ILM flap with no gas tamponade technique. Patients will be instructed to avoid excessive movement and adopt a sit up/supine posture for the first 24 hours, beyond which there will be no posturing restriction.
  Interventions: Procedure: ILM flap with no gas tamponade

INTERVENTIONS:
Procedure: Conventional surgery — Pars plana vitrectomy (PPV) with temporal internal limiting membrane (ILM) flap would be performed. Perfluorocarbon liquid (PFCL) or viscoelastic may be used as an adjunct. Air/Fluid exchange would be performed at the end of surgery, further exchange of air with 8-14% octafluoropropane (C3F8) would be performed based on operating surgeon's discretion. In cases a temporal ILM flap could not be created, an ILM flap would be created from other quadrants, for example, a nasal ILM would be created instead. Patients with visually significant cataract may undergo concomitant phacoemulsification and intraocular lens implantation or deferred to post-operative month 6-12. Patients would be instructed to adopt a face-down posturing in the first 5 days following operation.
  Arms: Conventional surgery
Procedure: ILM flap with no gas tamponade — Pars plana vitrectomy with temporal internal limiting membrane (ILM) flap would be performed. The ILM flap would be stabilised over the macular hole using perfluorocarbon liquid (PFCL) followed by sub-PFCL dispersive viscoelastic injection. The PFCL would be removed towards the end of surgery. In cases a temporal ILM flap could not be created, an ILM flap would be created from other quadrants, for example, a nasal ILM would be created instead. Concomitant phacoemulsification and intraocular lens implantation would be performed in patients with visually significant cataract or deferred to post-operative month 6-12. Patients will be instructed to avoid excessive movement and adopt a face forward/ supine position for first 24 hours. Afterwards, there would be no restriction on post-operative posturing.
  Arms: Internal limiting membrane (ILM) flap with no gas tamponade

SUMMARY:
Full-thickness macular hole (MH) is a common sight threatening macular condition with a prevalence of 3.3 per 1000 individuals. Prompt surgical repair of MH is imperative in preventing irreversible vision loss from MH as the majority of patients would experience progressive loss of central vision, often resulting in visual acuity (VA) of 20/200 or worse and the spontaneous closure rate is less than 10%.

Pars plana vitrectomy (PPV) with internal limiting membrane (ILM) peeling (with or without ILM flap) and gas tamponade, herein referred to as conventional surgery, is the current standard-of-care surgical technique in repairing MH.

Recently, a novel surgical technique that omits the need of gas tamponade to repair MH has been proposed, early results from retrospective studies were encouraging.

The purpose of this prospective international multi-centre randomised controlled study is to compare the efficacy and safety of two surgical techniques in treating MH:

1. Conventional surgery: PPV with ILM peeling and gas or silicone oil tamponade
2. ILM flap with no gas tamponade surgery: PPV with ILM flap with no gas tamponade

DETAILED DESCRIPTION:
MH is a common macular condition that requires prompt surgical intervention to prevent irreversible vision loss. Conventional surgical repair of MH involves PPV, ILM peeling and gas tamponade followed by post-operative face down posturing. The use of gas tamponade, however, is associated with impairment of vision in the early post-operative period and restriction of air travel. Moreover, fluorinated ophthalmic gases are potent green house gases that contribute to global warming.

Recently, a novel surgical technique to repair MH without endotamponade has been proposed, termed the ILM flap with no gas tamponade technique.

There is currently no published randomised controlled trial comparing the efficacy and safety of MH repair using conventional surgical technique and the ILM flap with no gas tamponade technique.

Patients with confirmed full thickness MH on optical coherence tomography will be screened and invited to join the study. Written informed consent will be obtained. Baseline screening will be performed.

Recruited study participants will be randomly allocated to one of the two study groups:

1. Conventional surgery: Participants will undergo PPV, ILM peeling and gas tamponade to repair the MH. They would be instructed to adopt a face down posture for at least 5 days post-operatively.
2. ILM flap with no gas tamponade surgery: Participants will undergo PPV, ILM flap. No gas tampons would be required and there would be no restriction on post-operative posturing.

Participants will be instructed to attend post-operative follow up visits to undergo routine clinical examination, visual acuity checking and retinal imaging performed.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Presence of full thickness macular hole in one eye (defined as full thickness discontinuity of neuro-sensory retina at the macula on optical coherence tomography)
* Able to comply to post-operative posture
* VA ≥0.05 and ≤0.8

Exclusion Criteria:

* Fellow eye enrolled in the study
* Eyes that underwent previous macular surgery
* Presence of maculopathy other than macular hole, epi-retinal membrane or myopic maculopathy. For example, age-related macular degeneration, diabetic macular edema or pre-existing macular scar
* Axial length >/= 28mm or presence of significant myopic chorio-retinal atrophy involving the fovea
* Minimum linear diameter >/=800µm
* Presence of contraindications to intraocular gas, such as advanced glaucoma or uncontrolled glaucoma
* Significant macular puckering (Govetto staging ≥ stage 2)
* Patients who are unable to give informed consent
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Macular hole closure rate | 3 months
  The primary outcome is the macular hole closure rate without additional vitrectomy/macular surgery at post-operative month 3.
  Closure of macular hole is defined as the presence of continuous retinal tissue over the retinal pigment epithelium (RPE) without bare RPE exposed to vitreous cavity on optical coherence tomography (OCT).

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) in the study eye | 12 months
  Best corrected visual acuity will be checked using the Snellen visual acuity chart
Pattern of macular hole closure | 12 months
  The pattern of macular hole closure will be assessed on optical coherence tomography
Rate of foveal gliosis | 12 months
  Based on optical coherence tomography.
Patients reported visual function | 12 months
  The patient reported visual function will be assessed using the National Eye Institute 25-item visual function questionnaire (NEI VFQ-25).
  The score ranges from 0-100, with higher score indicating better visual function.
Vision Preference Value Scale | 12 months
  Using a previously validated questionnaire to determine vision preference value and treatment preferences.
  Preference values were graded on a scale from 0 to 1, with 0 indicating death and 1 indicating perfect health with perfect vision.
Metamorphosia score | 12 months
  Using M-CHARTS (Inami & Co., Ltd., Tokyo, Japan) Ranges from 0-10. 0 indicates no metamorphopsia and 10 indicates severe metamorphopsia.

OTHER OUTCOMES:
Number of participants with surgery related adverse events | 12 months
  Include all post-operative complications, such as endophthalmitis, retinal detachment, re-opening of macular hole, intraocular pressure spike and hypotony.
Retinal sensitivity | 12 months
  Microperimetry will be performed to assess the retinal sensitivity. This is an exploratory outcome and will be performed in selected patients only.

CONTACTS AND LOCATIONS:
Overall Officials: Simon KH Szeto, MBChB, FRCOphth, Principal Investigator — Department of Ophthalmology and Visual Sciences, The Chinese University of Hong Kong
Locations (3):
- Hong Kong Eye Hospital, Hong Kong, Hong Kong
- Poznan University of Medical Sicences, University Hospital in Poznan, Poznan, Poland
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wada I, Yoshida S, Kobayashi Y, Zhou Y, Ishikawa K, Nakao S, Hisatomi T, Ikeda Y, Ishibashi T, Sonoda KH. Quantifying metamorphopsia with M-CHARTS in patients with idiopathic macular hole. Clin Ophthalmol. 2017 Sep 20;11:1719-1726. doi: 10.2147/OPTH.S144981. eCollection 2017. PMID 29033537
- [Background] Linz MO, Bressler NM, Chaikitmongkol V, Sivaprasad S, Patikulsila D, Choovuthayakorn J, Watanachai N, Kunavisarut P, Menon D, Tadarati M, Delalibera Pacheco K, Sanyal A, Scott AW. Vision Preference Value Scale and Patient Preferences in Choosing Therapy for Symptomatic Vitreomacular Interface Abnormality. JAMA Ophthalmol. 2018 Jun 1;136(6):658-664. doi: 10.1001/jamaophthalmol.2018.1272. PMID 29800983
- [Background] Chan CW, Wong D, Lam CL, McGhee S, Lai WW. Development of a Chinese version of the National Eye Institute Visual Function Questionnaire (CHI-VFQ-25) as a tool to study patients with eye diseases in Hong Kong. Br J Ophthalmol. 2009 Nov;93(11):1431-6. doi: 10.1136/bjo.2009.158428. Epub 2009 Jun 9. PMID 19515645
- [Background] Stopa M, Ciesielski M, Rakowicz P. Macular Hole Closure Without Endotamponade Application. Retina. 2023 Apr 1;43(4):688-691. doi: 10.1097/IAE.0000000000002850. Epub 2020 May 25. PMID 32453068
- [Background] Szeto SKH, Yu AHY, Tsang CW, Mohamed S, Chen LJ, Lai TYY. COMPLEX MACULAR HOLE CLOSURE BY TEMPORAL INTERNAL LIMITING MEMBRANE FLAP WITHOUT ENDOTAMPONADE. Retina. 2024 Nov 1;44(11):1915-1922. doi: 10.1097/IAE.0000000000004201. PMID 39436300